CLINICAL TRIAL: NCT01980875
Title: A Phase 3, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Idelalisib in Combination With Obinutuzumab Compared to Chlorambucil in Combination With Obinutuzumab for Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Efficacy and Safety of Idelalisib in Combination With Obinutuzumab Compared to Chlorambucil in Combination With Obinutuzumab for Previously Untreated Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-312-0118; 2013-004551-20 (EudraCT Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Chlorambucil; obinutuzumab

STUDY DESIGN:
Intervention Model Description: Safety Run-In Phase: Single Group; Randomized Phase: Parallel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-In: Idelalisib+obinutuzumab (Experimental): Participants will receive idelalisib for 96 weeks and obinutuzumab over 21 weeks. Following 4 weeks of treatment, safety data will be reviewed by an independent data monitoring committee (DMC). If acceptable tolerability is observed, the randomized portion of the study will begin.
  Interventions: Drug: Idelalisib; Drug: Obinutuzumab
- Randomized: Idelalisib+obinutuzumab (Experimental): Participants will receive idelalisib for 96 weeks and obinutuzumab over 21 weeks.
  Interventions: Drug: Idelalisib; Drug: Obinutuzumab
- Randomized: Obinutuzumab+chlorambucil (Active Comparator): Participants will receive obinutuzumab over 21 weeks and chlorambucil over 23 weeks.
  Interventions: Drug: Chlorambucil; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Idelalisib — 150 mg tablet administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®
  Arms: Randomized: Idelalisib+obinutuzumab; Safety Run-In: Idelalisib+obinutuzumab
Drug: Chlorambucil — 2 mg tablets administered at a dose of 0.5 mg/kg orally every other week for a total of 12 doses
  Arms: Randomized: Obinutuzumab+chlorambucil
Drug: Obinutuzumab — 1000 mg/40 mL single-use vials administered intravenously for a total of 8 doses over 21 weeks

SUMMARY:
The primary objective of this study is to evaluate the effects of idelalisib with obinutuzumab versus the combination of chlorambucil and obinutuzumab on progression-free survival (PFS) in participants with previously untreated chronic lymphocytic leukemia (CLL).

An increased rate of deaths and serious adverse events (SAEs) among participants with front-line CLL and early-line indolent non-Hodgkin lymphoma (iNHL) treated with idelalisib in combination with standard therapies was observed by the independent data monitoring committee (DMC) during regular review of 3 Gilead Phase 3 studies. Gilead reviewed the unblinded data and terminated those studies in agreement with the DMC recommendation and in consultation with the US Food and Drug Administration (FDA). All front-line studies of idelalisib, including this study, were also terminated.

ELIGIBILITY:
Key Inclusion Criteria:

* Not a candidate for fludarabine therapy based on either:

  1. creatinine clearance < 70 mL/min, or
  2. Cumulative Illness Rating Scale score > 6, by assessment of the investigator
* Diagnosis of B-cell CLL, with diagnosis established according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL)
* No prior therapy for CLL other than corticosteroids for disease complications.
* CLL that warrants treatment
* Presence of measurable lymphadenopathy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Key Exclusion Criteria:

* Known histological transformation from CLL to an aggressive lymphoma (ie, Richter transformation)
* Known presence of myelodysplastic syndrome
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of randomization
* Ongoing liver injury
* Ongoing drug-induced pneumonitis
* Ongoing inflammatory bowel disease
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy other than corticosteroids
* Concurrent participation in another therapeutic clinical trial
* Undergone major surgery within 30 days prior to randomization
* Known hypersensitivity or intolerance to any of the active substances or excipients in the formulations for idelalisib, obinutuzumab, or chlorambucil
* History of non-infectious pneumonitis
* Received last dose of study drug on another therapeutic clinical trial within 30 days prior to randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- United States (6):
  - Sansum Clinic, Santa Barbara, California
  - UCLA Jonsson Comprehensive Cancer Center, Santa Monica, California
  - Innovative Clinical Research Institute, Whittier, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Gabrail Cancer Center Research, Canton, Ohio
  - Saint Francis Cancer Center, Greenville, South Carolina
- St Vincent Hospital, Sydney, Darlinghurst, New South Wales, Australia
- UZ Ghent- hematology, Ghent, Belgium
- Royal Victoria Regional Health Centre - Simcoe Musk, Barrie, Ontario, Canada
- France (2):
  - Centre Hospitalier du Mans, Le Mans
  - Centre Hospitalier de Perpignan, Perpignan
- Poland (5):
  - Szpital Specjalistyczny w Brzozowie, Oddzial Hematologii Onkologicznej, Brzozów, Podkarpackie Voivodeship
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Wojewódzki Szpital Specjalistyczny w Legnicy, Legnica
  - Wojewodzki Szpital Specjalistyczny, im. M. Kopernika Klinika Hematologii Uniwersytetu Medycznego, Lodz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych z Warminsko-Mazurskim Centrum Onkologii w Olsztynie Oddzial Hematologii, Olsztyn
- Hospital Universitario de Salamanca, Salamanca, Spain
- East Kent Hospitals University NHS Foundation Trust, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe, and North America. The first participant was screened on 21 April 2015. The last study visit occurred on 13 May 2016.
Pre-assignment Details: 80 participants were screened.
Groups:
- Safety Run-In: Idelalisib+Obinutuzumab: Idelalisib (Zydelig®) 150 mg tablet twice daily + obinutuzumab 1000 mg/40 mL intravenously for a total of 8 doses over 21 weeks
- Randomized: Idelalisib+Obinutuzumab: Idelalisib 150 mg tablet twice daily + obinutuzumab 1000 mg/40 mL intravenously for a total of 8 doses over 21 weeks
- Randomized: Obinutuzumab+Chlorambucil: Chlorambucil 0.5 mg/kg, as 2 mg tablets every other week for a total of 12 doses + obinutuzumab 1000 mg/40 mL intravenously for a total of 8 doses over 21 weeks
Period: Overall Study
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Started | 8 | 25 | 24
Completed | 0 | 0 | 0
Not Completed | 8 | 25 | 24
Not completed — Withdrew Consent | 1 | 1 | 1
Not completed — Study Terminated by Sponsor | 7 | 24 | 22
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis Set: participants who were randomized regardless of whether participants received any study drug(s), or received a different regimen from the regimen to which they were randomized.
Groups:
- Safety Run-In: Idelalisib+Obinutuzumab; Randomized: Idelalisib+Obinutuzumab: Idelalisib 150 mg tablet twice daily + obinutuzumab 1000 mg/40 mL intravenously for a total of 8 doses over 21 weeks
- Total: Total of all reporting groups
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil | Total
Number analyzed (Participants) | 8 | 25 | 24 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.10) | 72.2 (8.23) | 71.1 (6.84) | 71.1 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 9 | 20
  Male | 5 | 17 | 15 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 0 | 1
  White | 7 | 22 | 21 | 50
  Other | 0 | 1 | 0 | 1
  Not Permitted | 0 | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 0 | 2
  Belgium | 0 | 1 | 1 | 2
  United States | 5 | 3 | 4 | 12
  Poland | 2 | 14 | 12 | 28
  United Kingdom | 0 | 1 | 2 | 3
  France | 0 | 3 | 2 | 5
  Australia | 0 | 1 | 3 | 4
  Spain | 0 | 1 | 0 | 1
Rai Stage [Count of Participants; unit: Participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL) with higher stages reflecting increasing severity.
  Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis with lymphadenopathy, Rai Stage II: Lymphocytosis with hepatomegaly or splenomegaly, Rai Stage III: Lymphocytosis with anemia, Rai Stage IV: Lymphocytosis with thrombocytopenia.
  Participants
    Stage I-II | 3 | 11 | 9 | 23
    Stage III-IV | 5 | 14 | 15 | 34
IgHV Mutation [Count of Participants; unit: Participants] — The mutation status of the unique immunoglobulin gene (IgHV) rearrangement in the monoclonal proliferation of B-cells in CLL can be used to predict aggressiveness of the disease. Participants with a mutated IgHV gene usually have a less aggressive and more indolent disease, with longer overall survival. Participants with an unmutated IgHV gene usually have a more aggressive disease and shorter overall survival.
  Participants
    Unmutated | 5 | 16 | 17 | 38
    Mutated | 3 | 9 | 7 | 19
17p Deletion in CLL Cells [Count of Participants; unit: Participants] — Participants with CLL who have deletion of 17p, a portion of the chromosome that acts to suppress cancer growth and is a recognized negative prognostic risk factor.
  Participants
    Present | 0 | 3 | 3 | 6
    Absent | 8 | 22 | 21 | 51

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) is defined as the interval from randomization to the first documentation of definitive disease progression or death from any cause. Definitive disease progression is CLL progression based on standard criteria, excluding lymphocytosis alone. PFS was to be assessed by an independent review committee (IRC).
Time Frame: Up to 11 months
Population: The study was terminated in agreement with the FDA due to urgent safety measures. Complete data were not collected for any participant.
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined as the proportion of participants who achieve a confirmed complete or partial response. ORR was to be assessed by an IRC.
Time Frame: Up to 11 months
Population: as for outcome 1
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Nodal Response Rate
Description: Nodal response rate is defined as the proportion of participants who achieve a 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters of index lesions. Nodal response rate was to be assessed by an IRC.
Time Frame: Up to 11 months
Population: as for outcome 1
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Complete Response Rate
Description: Complete response rate is defined as the proportion of participants who achieve a confirmed complete response. Complete response rate was to be assessed by an IRC.
Time Frame: Up to 11 months
Population: as for outcome 1
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval from randomization to death from any cause. Overall survival was to be assessed by an IRC.
Time Frame: Up to 11 months
Population: as for outcome 1
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Minimal Residual Disease Negativity Rate at Week 36
Description: Minimal residual disease (MRD) negativity rate is defined as the proportion of participants with MRD < 10^-4 assessed by flow cytometry in bone marrow at Week 36 after therapy initiation. For participants receiving the final dose of obinutuzumab after the original scheduled date, the MRD assessment was performed no less than 12 weeks after the last dose of obinutuzumab. MRD negativity rate was to be assessed by an IRC.
Time Frame: Up to 11 months
Population: as for outcome 1
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum: 12 months)
Description: Safety Analysis Set: participants who received at least 1 dose of study drug, with treatment group designated according to actual treatment received
Arm/Group | Safety Run-In: Idelalisib+Obinutuzumab | Randomized: Idelalisib+Obinutuzumab | Randomized: Obinutuzumab+Chlorambucil
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/8 | 12/24 | 8/23
Other Adverse Events (participants affected / at risk) | 8/8 | 19/24 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-In: Idelalisib+Obinutuzumab (N=8) | Randomized: Idelalisib+Obinutuzumab (N=24) | Randomized: Obinutuzumab+Chlorambucil (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Secondary immunodeficiency (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-In: Idelalisib+Obinutuzumab (N=8) | Randomized: Idelalisib+Obinutuzumab (N=24) | Randomized: Obinutuzumab+Chlorambucil (N=23)
Anaemia (Blood and lymphatic system disorders) | 2 | 6 | 2
Neutropenia (Blood and lymphatic system disorders) | 4 | 6 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 1
Dry eye (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 2 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 2
Influenza like illness (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 1
Pyrexia (General disorders) | 1 | 1 | 4
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 3 | 14
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 7 | 5 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 5 | 1
Blood creatinine increased (Investigations) | 0 | 2 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0 | 0
Circadian rhythm sleep disorder (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2
Psychomotor skills impaired (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 0
Restlessness (Psychiatric disorders) | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was terminated in agreement with the FDA due to urgent safety measures. Complete data were not collected for any participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years